CLINICAL TRIAL: NCT00616967
Title: A Multi-Institutional Double-Blind Phase II Study Evaluating Response and Surrogate Biomarkers to Carboplatin and Nab-Paclitaxel (CP) With or Without Vorinostat as Preoperative Chemotherapy in HER2-negative Primary Operable Breast Cancer
Brief Title: Carboplatin and Nab-Paclitaxel With or Without Vorinostat in Treating Women With Newly Diagnosed Operable Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: J0785; P30CA006973 (NIH); NA_00012756 (Other: JHM IRB); JHOC-SKCCC-J0785 (Other: SKCCC at Johns Hopkins); JHOC-J0785 (Other: SKCCC at Johns Hopkins); CDR0000586335 (Other: other)
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; ductal breast carcinoma; lobular breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Lobular | interventions — Carboplatin; Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Vorinostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Active Comparator): Patients receive carboplatin IV and paclitaxel albumin-stabilized nanoparticle formulation IV on day 1 and an oral placebo on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Other: placebo
- Arm II (Experimental): Patients receive carboplatin and paclitaxel albumin-stabilized nanoparticle formulation as in arm I and oral vorinostat on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Drug: vorinostat

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Paraplatin
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV
  Other Names: Abraxane, nab-Paclitaxel
Drug: vorinostat — Given orally
  Other Names: Zolinza
  Arms: Arm II
Other: placebo — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Vorinostat may also help carboplatin and paclitaxel albumin-stabilized nanoparticle formulation work better by making tumor cells more sensitive to the drugs. Giving chemotherapy with or without vorinostat before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This randomized phase II trial is studying how well giving carboplatin together with paclitaxel albumin-stabilized nanoparticle formulation works with or without vorinostat in treating women with breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine pathological complete response (pCR) rates in patients with HER2-negative primary operable breast cancer treated with neoadjuvant therapy comprising carboplatin and paclitaxel albumin-stabilized nanoparticle formulation (CP) with vs without vorinostat.

Secondary

* To evaluate the safety of these regimens in these patients.
* To estimate clinical complete response (cCR) rates in patients treated with these regimens.
* To correlate baseline and change (day 15) in surrogate uptake values (SUV) on FDG-PET with pathological and clinical response in patients treated with these regimens, and to determine what percent of women with ≥ 25% or ≥ 50% reduction in SUV on day 15 achieve a pCR and a cCR to CP with vs without vorinostat.
* To correlate baseline and change in markers of proliferation with pathological and clinical response in patients treated with these regimens.
* To evaluate long term outcomes (e.g., recurrence of the breast cancer, development of a new cancer, or death) for patients treated with these regimens.

Tertiary

* To evaluate baseline and change in candidate gene methylation and expression profiles.
* To evaluate baseline and change in tissue and peripheral blood mononuclear cell histone acetylation.
* To compare cCR and pCR in women with basal-like features versus other subtypes.

OUTLINE: This is a multicenter, randomized, double-blind, phase II study (primary study portion) with a 6-12 patient run-in portion.

* Run-in portion: Patients receive carboplatin IV and paclitaxel albumin-stabilized nanoparticle formulation IV on day 1 and oral vorinostat on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity. Once safety of the combination of chemotherapy and vorinostat is confirmed, subsequently enrolled patients are entered to the primary study portion.
* Primary study portion: Patients are stratified by hormone receptor status (estrogen receptor [ER]-negative and progesterone receptor [PR]-negative vs ER-positive and/or PR-positive). Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive carboplatin IV and paclitaxel albumin-stabilized nanoparticle formulation IV on day 1 and an oral placebo on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive carboplatin and paclitaxel albumin-stabilized nanoparticle formulation as in arm I and oral vorinostat on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.

Within 2-4 weeks after completion of neoadjuvant chemotherapy, patients undergo breast conserving surgery or mastectomy at the discretion of the treating physician.

Patients undergo tumor tissue biopsy at baseline, day 15, and at the time of definitive surgery. Samples are analyzed by immunohistochemistry (IHC), RNA extraction, and gene expression analysis using RT-PCR to identify candidate markers for response and molecular profiles that may be relevant to an understanding of drug mechanisms. Methylation of relevant genes (e.g., ERalpha, APC-1, RARbeta, cyclin D2, Twist, RASSF1A, and HIN-1) are evaluated by quantitative multiplex methylation-specific PCR. Changes in gene expression as a result of treatment are determined by IHC or quantitative RT-PCR. Blood samples are collected at baseline, day 15, at the time of definitive surgery, and 4 weeks after surgery for DNA methylation studies, pharmacogenomic studies, and histone acetylation assays. Patients also undergo fludeoxyglucose F 18-positron emission tomography (FDG-PET) or PET/CT at baseline and day 15 to assess treatment response as measured by standardized uptake values.

After completion of study treatment, patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed infiltrating ductal breast cancer by core needle biopsy

  * Mixed ductal and lobular disease allowed
  * Infiltrating lobular cancer allowed in the run-in portion only
* Unresected, clinically measurable disease, meeting 1 of the following clinical staging criteria:

  * T2, T3, or T4 lesion, any N, M0
  * T1c, N1-3,M0
* Patients with skin metastases to the ipsilateral breast for whom chemotherapy is planned prior to definitive surgery are eligible for the primary study portion
* HER2-negative disease
* Hormone receptor status* meeting 1 of the following criteria:

  * Estrogen receptor (ER)-negative and progesterone receptor (PR)-negative
  * ER-positive (grade II or III) and PR-positive or PR-negative NOTE: *Any ER or PR status for the run-in portion

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Menopausal status not specified
* ANC ≥ 1,500/mm³
* Platelet count ≥ 150,000/mm³
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 times the upper limit of normal (ULN)
* Creatinine clearance ≥ 50 mL/min
* Total bilirubin normal
* AST(SGOT) and ALT(SGPT) ≤ 2.5 times (ULN)
* alkaline phosphatase ≤ 2.5 times ULN
* PT such that INR ≤ 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and PTT ≤ ULN
* Adequate cardiac function defined as no evidence of PR prolongation or AV block on baseline electrocardiogram (ECG)
* Willing to use effective, non-hormonal contraception while on treatment and for at least 3 months thereafter
* Not pregnant or nursing
* No pre-existing peripheral neuropathy ≥ grade 2
* No history of severe hypersensitivity reaction to any drug formulated with polysorbate 80 or to E. coli-derived products
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat
* No medical condition which, in the opinion of the investigator, puts the patient at risk of potentially serious complications while on this therapy

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior valproic acid or other histone deacetylase inhibitor
* No prior chemotherapy, radiotherapy, or endocrine therapy for this cancer

  * Prior tamoxifen or raloxifene or another agent for prevention of breast cancer allowed as long as the patient has discontinued the treatment ≥ 1 month prior to baseline study biopsy
* No systemic treatment for prior cancer within the past 5 years (primary study portion)
* No prior or ongoing systemic treatment for this cancer (primary study portion)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent histone deacetylase inhibitor
* No other concurrent chemotherapy, antiestrogen therapy, radiotherapy, or other investigational systemic therapy
* No other concurrent biologic therapy
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-05; Primary Completion 2014-06 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (5):
- United States (5):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Indiana University Purdue University of Indianapolis, Indianapolis, Indiana
  - Anne Arundel Health System, Annapolis, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic Cancer Center, Rochester, Minnesota

REFERENCES:
- [Result] Connolly RM, Leal JP, Goetz MP, Zhang Z, Zhou XC, Jacobs LK, Mhlanga J, O JH, Carpenter J, Storniolo AM, Watkins S, Fetting JH, Miller RS, Sideras K, Jeter SC, Walsh B, Powers P, Zorzi J, Boughey JC, Davidson NE, Carey LA, Wolff AC, Khouri N, Gabrielson E, Wahl RL, Stearns V. TBCRC 008: early change in 18F-FDG uptake on PET predicts response to preoperative systemic therapy in human epidermal growth factor receptor 2-negative primary operable breast cancer. J Nucl Med. 2015 Jan;56(1):31-7. doi: 10.2967/jnumed.114.144741. Epub 2014 Dec 4. PMID 25476537
- [Result] Connolly RM, Fackler MJ, Zhang Z, Zhou XC, Goetz MP, Boughey JC, Walsh B, Carpenter JT, Storniolo AM, Watkins SP, Gabrielson EW, Stearns V, Sukumar S. Tumor and serum DNA methylation in women receiving preoperative chemotherapy with or without vorinostat in TBCRC008. Breast Cancer Res Treat. 2018 Jan;167(1):107-116. doi: 10.1007/s10549-017-4503-2. Epub 2017 Sep 16. PMID 28918548

RESULTS

PARTICIPANT FLOW:
Groups:
- Run-in Phase (Arm 0): Phase 0 - To confirm safety and dosing prior to moving to randomized phase 2 portion (Arms 1 and 2).
  Patients receive carboplatin and paclitaxel albumin-stabilized nanoparticle formulation as in arm I and oral vorinostat on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  carboplatin: Given IV paclitaxel albumin-stabilized nanoparticle formulation: Given IV vorinostat: Given orally
- Placebo (Arm I): Patients receive carboplatin IV and paclitaxel albumin-stabilized nanoparticle formulation IV on day 1 and an oral placebo on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  carboplatin: Given IV
  paclitaxel albumin-stabilized nanoparticle formulation: Given IV
  placebo: Given orally
- Vorinostat (Arm II): Patients receive carboplatin and paclitaxel albumin-stabilized nanoparticle formulation as in arm I and oral vorinostat on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  carboplatin: Given IV
  paclitaxel albumin-stabilized nanoparticle formulation: Given IV
  vorinostat: Given orally
Period: Overall Study
Arm/Group | Run-in Phase (Arm 0) | Placebo (Arm I) | Vorinostat (Arm II)
Started | 6 | 31 | 31
Completed | 6 | 31 | 30
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The information for the primary populations for analysis are included (Placebo and Vorinostat arms). The initial "run-in phase" of 6 participants was conducted to confirm safety and dosing for the combination of vorinostat with chemotherapy only, and these data are not a part of our primary study analyses.
Groups:
- Placebo (Arm 1): Patients receive carboplatin IV and paclitaxel albumin-stabilized nanoparticle formulation IV on day 1 and an oral placebo on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  carboplatin: Given IV
  paclitaxel albumin-stabilized nanoparticle formulation: Given IV
  placebo: Given orally
- Vorinostat (Arm 2): Patients receive carboplatin and paclitaxel albumin-stabilized nanoparticle formulation as in arm I and oral vorinostat on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  carboplatin: Given IV
  paclitaxel albumin-stabilized nanoparticle formulation: Given IV
  vorinostat: Given orally
- Total: Total of all reporting groups
Arm/Group | Placebo (Arm 1) | Vorinostat (Arm 2) | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Median (Full Range); unit: years] | 48 [24 to 72] | 48 [31 to 68] | 48 [24 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 19 | 24 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 31 | 62
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG (Eastern Cooperative Oncology Group) criteria is a measure of patient performance status due to symptoms. A score of ECOG = 0 is defined as a person who is asymptomatic. A score of ECOG =1 is a defined as a person who has symptoms, but is fully ambulatory.
  Participants
    ECOG 0 | 30 | 29 | 59
    ECOG 1 | 1 | 2 | 3
Tumor Size [Median (Full Range); unit: centimeters] | 5 [1.7 to 18] | 4 [1.5 to 11.5] | 4 [1.5 to 18]
Nodal Status [Count of Participants; unit: Participants]
  Negative | 10 | 14 | 24
  Positive | 21 | 17 | 38
Tumor Grade [Count of Participants; unit: Participants] — Tumor grade is the description of a tumor based on how abnormal the tumor cells and tissue look under a microscope. It is an indicator of how quickly a tumor is likely to grow and spread. If the cells of the tumor are close to those of normal cells, the tumor is called "well-differentiated." Tumors that are "undifferentiated" or "poorly differentiated" have abnormal-looking cells and may lack normal tissue structures. A grade = 1 means well differentiated (low grade). A grade = 2 means moderately differentiated (intermediate grade). A grade = 3 means poorly differentiated (high grade).
  Participants
    Grade 2 | 11 | 7 | 18
    Grade 3 | 20 | 24 | 44
Receptor Status [Count of Participants; unit: Participants] — Estrogen receptors (ER) and Progesterone receptors (PR) are found in breast cancer cells that depend on estrogen and related hormones to grow. If breast cancer cells have estrogen receptors, the cancer is called ER-positive breast cancer (ER+) . If breast cancer cells have progesterone receptors, the cancer is called PR-positive breast cancer (PR+). If the cells do not have either of these two receptors, the cancer is called ER/PR-negative (ER- and PR-).
  Participants
    ER-/PR- | 12 | 12 | 24
    ER+/PR+ | 12 | 10 | 22
    ER+/PR- | 6 | 6 | 12
    ER-/PR+ | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate
Description: The primary end point was pCR, defined as no viable invasive cancer in breast and axilla. All other cases were defined as non-pCR. The pCR rate was determined in each arm separately by performing an intent-to-treat (ITT) analysis of all randomized patients. Patients with unknown pCR status were considered non-responders. Computation of associated 90% confidence intervals did not account for the sequential design.
Time Frame: Time of breast cancer surgery
Population: The information for the primary populations for analysis are included (Placebo and Vorinostat arms). Data for this outcome measure was not collected from the initial "run-in phase" of 6 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 31 | 31
Participants | 9 | 8
Statistical Analysis 1: Comparison: Arm I vs Arm II; Patients were stratified by hormone receptor status and randomly assigned to either arm 1 or 2. This study was designed using Simon's two-stage design for each arm in parallel. Interim analysis of early stopping for futility was conducted for the first 32 patients (16 patients per arm) and the study proceeded as more than 2 patients achieved a pCR in each arm (31 patients per arm). This design had 80% power to detect a 25% pCR rate versus a null rate of 10% with a type I error rate of 0.10; Test type: Superiority or Other; Pathological complete response rate = 0.274, 95% CI 2-sided [0.169 to 0.402] — The Estimation Parameter provided above is for overall pCR for both arms combined. We estimated pCR for each arm separately as well
Statistical Analysis 2: Comparison: Arm I; Test type: Superiority or Other; pCR in placebo arm (arm 1) = 0.29, 95% CI 2-sided [0.142 to 0.48]
Statistical Analysis 3: Comparison: Arm II; Test type: Superiority or Other; pCR in vorinostat arm (arm 2) = 0.258, 95% CI 2-sided [0.119 to 0.446]

2. Secondary Outcome: Safety as Measured by Number of Participants Who Experience Adverse Events
Description: Number of participants who experience adverse events as defined by NCI CTCAE version 3.0
Time Frame: up to 30 days post-treatment
Measure: Count of Participants; unit: Participants
Groups:
- Run-in Phase (Arm 0): Patients receive carboplatin and paclitaxel albumin-stabilized nanoparticle formulation and oral vorinostat on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  carboplatin: Given IV
  paclitaxel albumin-stabilized nanoparticle formulation: Given IV
  vorinostat: Given orally
Arm/Group | Run-in Phase (Arm 0) | Placebo (Arm 1) | Vorinostat (Arm 2)
Number analyzed (Participants) | 6 | 31 | 31
Participants | 6 | 31 | 31

3. Secondary Outcome: Number of Participants With Clinical Complete Response (cCR)
Description: cCR in the breast on physical is defined as the absence of any palpable abnormality on breast exam Iie: no skin or breast thickening, mass or associated skin or nipple changes)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Arm I) | Vorinostat (Arm II)
Number analyzed (Participants) | 31 | 31
Participants | 16 | 15

4. Secondary Outcome: Change in Standard Uptake Value (SULmax) From Baseline to Day 15 on FDG-PET
Description: Change in standard uptake value (SULmax) as measured by percentage reduction of SULmax. The standard uptake value used for the PET analysis was SULmax, which is the standard uptake value normalized for lean body mass.
Time Frame: Baseline and day 15
Population: 16/17 "Responders" (from Outcome 1) had PET data evaluable for analysis; 43/45 "non-responders" (from Outcome 1) had PET data evaluable for analysis. Reasons for PET data not evaluable included technically invalid 18F-FDG PET data (2 participants) and no available Day 15 18F-FDG PET data (1 participant).
Measure: Median (Full Range); unit: percentage reduction in SULmax
Groups:
- Responders: Pooled data from participants who received a pathologic complete response across arms.
- Non-Responders: Pooled data from participants who did not receive a pathologic complete response across arms.
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 16 | 43
percentage reduction in SULmax | 63 [4.4 to 85.3] | 32.9 [-84.2 to 77.1]
Statistical Analysis 1: Comparison: Responders vs Non-Responders; The estimates provided are based upon a multivariate analysis using a logistic regression adjusting for hormone receptor status. Patients with ≥50% reduction in SULmax were more likely to achieve a pCR; Test type: Superiority or Other; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 5.1, 95% CI 2-sided [1.3 to 22.7]

5. Secondary Outcome: Absolute Change From Baseline in Ki-67
Time Frame: Change from baseline to Cycle 1-Day 15
Population: Only 8/17 and 36/45 specimens were evaluable for Ki-67 at both baseline and Day 15. Nonevaluable samples had no tumor cells present or Ki-67 unavailable at either or both time points.
Measure: Mean (Standard Deviation); unit: percent change in Ki-67
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 8 | 36
percent change in Ki-67 | 7.0 (15.8) | 12.0 (22.7)

6. Secondary Outcome: Change in Cumulative Methylation Index (CMI)
Description: Change of CMI from baseline to Day 15 (D15), defined as log(D15 CMI + 1/baseline CMI + 1). The CMI was calculated as a sum of all gene-specific methylation indexes within a panel of 10 genes which included: HIST1H3C, AKR1B1, GPX7, HOXB4, TMEFF2, RASGRF2, COL6A2, ARHGEF7, TM6SF1, and RASSF1A.
Time Frame: Change from baseline to Day 15
Population: Methylation data was only evaluable in participants with both baseline and D15 tissue (48/62) and serum (58/62) specimens.
Measure: Median (Full Range); unit: CMI
Groups:
- Combined Arm I and Arm II: Tissue and serum samples from all participants in the actual study (combination of both arms).
Arm/Group | Combined Arm I and Arm II
Number analyzed (Participants) | 62
CMI
  Tissue CMI change from baseline: number analyzed (Participants) | 48
  Tissue CMI change from baseline | 14 [-310 to 69]
  Serum CMI change from baseline: number analyzed (Participants) | 58
  Serum CMI change from baseline | 0 [-120 to 29]

7. Secondary Outcome: Cumulative Methylation Index (CMI) at Day 15
Time Frame: Day 15
Population: Methylation data was only evaluable in 11/17 and 39/45 participants.
Measure: Median (Full Range); unit: CMI
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 11 | 39
CMI | 10 [1 to 40] | 44 [0 to 163]

8. Secondary Outcome: Number of Participants Who Experience Death During Treatment
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Phase (Arm 0) | Placebo (Arm I) | Vorinostat (Arm II)
Number analyzed (Participants) | 6 | 31 | 31
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Who Develop New Cancer
Time Frame: Up to death of last participant (duration unknown)
Reporting Status: Not Posted

10. Secondary Outcome: Number of Participants With Recurrence of Breast Cancer
Time Frame: Up to death of last participant (duration unknown)
Reporting Status: Not Posted

11. Secondary Outcome: Overall Survival
Time Frame: Up to death of last participant (duration unknown)
Reporting Status: Not Posted

12. Post Hoc Outcome: Baseline and Change in Continuous Variables (e.g., Candidate Gene Methylation, Expression Profiles, Tissue, and Peripheral Blood Mononuclear Cell Histone Acetylation)
Time Frame: Time of breast cancer surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days following the 12 weeks of treatment
Groups:
- Run-in Phase (Arm 0): Phase 0 - To confirm safety and dosing prior to moving to randomized phase 2 portion (Arms 1 and 2).
  Patients receive carboplatin and paclitaxel albumin-stabilized nanoparticle formulation as in arm I and oral vorinostat on days 1-3. Treatment repeats weekly for 12 weeks in the absence of disease progression or unacceptable toxicity.
  carboplatin: Given IV
  paclitaxel albumin-stabilized nanoparticle formulation: Given IV
  vorinostat: Given orally
  Events summarized in this arm are those that met 5% reporting threshold in Arms I and II.
Arm/Group | Run-in Phase (Arm 0) | Arm I | Arm II
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/6 | 3/31 | 1/31
Other Adverse Events (participants affected / at risk) | 6/6 | 31/31 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Phase (Arm 0) (N=6) | Arm I (N=31) | Arm II (N=31)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Phase (Arm 0) (N=6) | Arm I (N=31) | Arm II (N=31)
Allergic reaction (Immune system disorders) | 0 (0) | 10 (10) | 1 (1)
Amemia (hemoglobin) (Blood and lymphatic system disorders) | 3 (3) | 9 (9) | 20 (20)
Neutropenia (neutrophils) (Blood and lymphatic system disorders) | 6 (6) | 28 (28) | 29 (29)
Thrombocytopenia (platelets) (Blood and lymphatic system disorders) | 1 (1) | 10 (10) | 15 (15)
ALT (elevated) (Investigations) | 0 (0) | 4 (4) | 1 (1)
Chills (General disorders) | 1 (1) | 4 (4) | 5 (5)
Fatigue (Gastrointestinal disorders) | 6 (6) | 31 (31) | 27 (27)
Insomnia (Psychiatric disorders) | 2 (2) | 6 (6) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 31 (31) | 29 (29)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (8) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (9) | 9 (9)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 17 (17) | 19 (19)
Constipation (Gastrointestinal disorders) | 2 (2) | 14 (14) | 18 (18)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 18 (18) | 18 (18)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 2 (2) | 6 (6)
Flatulence (Gastrointestinal disorders) | 1 (1) | 7 (7) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 9 (9) | 7 (7)
Mucositis (Gastrointestinal disorders) | 3 (3) | 10 (10) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 25 (25) | 29 (29)
Taste alteration (Gastrointestinal disorders) | 5 (5) | 13 (13) | 17 (17)
Vomiting (Gastrointestinal disorders) | 2 (2) | 10 (10) | 19 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 14 (14) | 5 (5)
Hot flashes (Vascular disorders) | 3 (3) | 8 (8) | 7 (7)
Upper respiratory infection (Infections and infestations) | 0 (0) | 10 (10) | 7 (7) — Sinus infection
Dizziness (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6) | 25 (25) | 20 (20)
Vision changes (Eye disorders) | 0 (0) | 4 (4) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 13 (13) | 15 (15)
Headache (Nervous system disorders) | 3 (3) | 8 (8) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 11 (11) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 0 (0)

LIMITATIONS AND CAVEATS:
A proportion of women received additional preoperative chemotherapy after study treatment,complicating the evaluation of primary endpoint and role of FDG-PET in predicting response. Limited matched samples for Ki67 analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No